CLINICAL TRIAL: NCT01398241
Title: Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of RO5267683 in an Adaptive, Randomized, Investigator-blind and Subject-blind, Multiple-ascending Dose, Placebo-controlled, Study Following Oral Administrations in Healthy Subjects for 28 Days
Brief Title: A Study of RO5267683 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP25214; 2011-000600-17 (EudraCT Number)
Record Dates: First submitted 2011-07-14; First posted 2011-07-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active (Experimental)
  Interventions: Drug: RO5267683
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: RO5267683 — Multiple ascending doses
  Arms: Active
Drug: placebo — Multiple ascending doses
  Arms: Placebo

SUMMARY:
This investigator-blind, subject-blind, randomized, placebo-controlled study will evaluate the safety, pharmacokinetics and pharmacodynamics of multiple ascending doses of RO5267683 in healthy volunteers. Subjects will be randomized to receive either RO5267683 or placebo orally daily for 28 days. Follow-up will be 10 weeks after the last dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects, 18 to 45 years of age,
* Body mass index (BMI) 18 to 30 kg/m2 inclusive, and a minimum weight of 50 kg at screening
* Female subjects must be surgically sterile or post-menopausal
* Male subjects must use a barrier method of contraception for the duration of the study and for 90 days after the last dose

Exclusion Criteria:

* History or evidence of any clinically significant disease or disorder
* Administration of an investigational drug or device within 3 months prior to dosing on Day 1
* Positive for hepatitis B, hepatitis C or HIV at screening
* Subjects on hormone replacement therapy who have not been receiving a stable dose for at least 2 months prior to start of dosing

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | 14 weeks

SECONDARY OUTCOMES:
Pharmacokinetics: Plasma concentrations | 14 weeks
Pharmacokinetics: Urine concentrations | 4 weeks
Lipid levels in the blood | 14 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Strasbourg, France